CLINICAL TRIAL: NCT04917926
Title: Effectiveness of Behavioural Economics-based Incentives on Glycaemic Control and Lifestyle in Adults With Newly Diagnosed Type 2 Diabetes: a Randomised Control Trial
Brief Title: Behavioural Economics-based Incentives in Adults With Type 2 Diabetes (BET2)
Acronym: BET2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BET2-v4-202106
Record Dates: First submitted 2021-04-28; First posted 2021-06-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Financial and social intervention (Experimental): Participants will receive the usual standard care (same as control group), loss-framed financial incentives, social incentives and weekly feedback on performance for 6 months.
  Interventions: Behavioral: Financial and social incentives
- Control (No Intervention): Participants will receive standard care including patient screening and education on diet, physical activity, and smoking conducted by a multi-disciplinary team. Participants in the control group will neither be told their baseline step count nor receive any feedback messages.
- Financial intervention (Experimental): Participants will receive the usual standard care (same as control group), loss-framed financial incentives, and weekly feedback on performance for 6 months.
  Interventions: Behavioral: Financial incentives

INTERVENTIONS:
Behavioral: Financial and social incentives — Participants will be credited with HK$1,000 in their virtual accounts at the beginning of the trial. After baseline step counts are gathered in the second week, they will lose HK$40 for each subsequent week that they do not meet their personal weekly step target. Regarding social incentives, participants will be placed in teams of six, receiving feedback of their physical activity performance, rankings within their groups, and positive messages for encouragement. Nominated supporters will be informed of participants' performance for social support.
  Arms: Financial and social intervention
Behavioral: Financial incentives — Participants will be credited with HK$1,000 in their virtual accounts at the beginning of the trial. After baseline step counts are gathered in the second week, they will lose HK$40 for each subsequent week that they do not meet their personal weekly step target.
  Arms: Financial intervention

SUMMARY:
A randomised control trial of adults with newly diagnosed type 2 diabetes to assess the effectiveness of behavioural economics-based incentives on healthy lifestyle behaviour, using a pragmatic trial approach.

DETAILED DESCRIPTION:
This is a randomised control trial of adults aged 30-70 with newly diagnosed type 2 diabetes within a year in Hong Kong to compare the effectiveness of financial incentives and combined financial and social incentives against a control group receiving standard care. We plan to recruit 261 participants and follow them for 9-months (6-month intervention period and a 3-month post-intervention follow-up period) to assess glycemic control and other health indicators. Participants will be randomly assigned to one of three groups (in ratio 1:1:1): arm A (financial incentives in addition to standard care), arm B (financial and social incentives in addition to standard care), and arm C (control arm receiving standard care). Financial incentives will be framed around loss aversion and the endowment effect. Social incentives will include peer competition, and social support. Financial and social incentives are to encourage increased physical activity and participants will use a pedometer to track activity. Participants are followed for an additional 3-months after the cessation of incentives to assess the sustainability of lifestyle changes.

This trial adopts a pragmatic study design based on the PRECIS-2 tool and RE-AIM frameworks.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults aged 30-70 years
* Capable of providing informed consent
* Resident in Hong Kong
* Able to communicate in English or Chinese
* Diagnosed with type 2 diabetes within past year
* 6.5% ≤ HbA1c ≤ 9.0%
* Willing to take blood tests
* Access to a phone to track physical activity and receive text messages
* Physically mobile for duration of the trial

Exclusion Criteria:

* Planned surgery in the next 6 months
* Biological impairment or health condition affecting the ability to walk, such as blindness, physical immobility, and paralysis
* Pregnant or breastfeeding
* On insulin for diabetes control

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | Baseline, 6-months, and 9-months
  The change in HbA1c levels

SECONDARY OUTCOMES:
Diabetes control | Baseline, 6-months, and 9-months
  Proportion of participants with good/excellent diabetes control (HbA1c threshold ≤ 7% & ≤ 6.5%)
Body weight control | Baseline, 6-months, and 9-months
  Change in body weight in kilograms; weight and height will be combined to report BMI in kg/m^2
Changes in lipid profile | Baseline, 6-months, and 9-months
  Changes in Total, HDL- and LDL-cholesterol, and Triglycerides
Change in blood pressure | Baseline, 6-months, and 9-months
  Assessed by the change in systolic and diastolic blood pressure
Glycaemic control | 6-months and 9-months
  Proportion of participants requiring an initiation of medication in diabetes management
Glycaemic control (addition of medications) | 6-months and 9-months
  Proportion of participants requiring an addition of medication(s) or increase in drug dosage in diabetes management
Walking performance | Weekly
  Assessed by proportion of participants meeting their daily step counts every week
Level of physical activity | Baseline, 6-months and 9-months
  Assessed by the structured and validated International Physical Activity Questionnaires (IPAQ); Both walking performance (Outcome 6) and the IPAQ score can be used for assessing the level of physical activity of participants

OTHER OUTCOMES:
Frequency of health service utilisation | Baseline, 6-months, and 9-months
  Number of medical appointment attendances and hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Jianchao Quan, MPH, BM BCh, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- School of Public Health, Li Ka Shing Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared in accordance with the University of Hong Kong Data Management Plan (DMP)
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available for at least 5 years after the release of publication of this study.
Access Criteria: Only data without personal information will be shared. The data will be shared for academic use only.
URL: https://hub.hku.hk/researchdata/staff2.htm